CLINICAL TRIAL: NCT00504816
Title: An Open Label, Single-sequence, Repeat-dose Study to Investigate the Effects of GSK189075 on the Pharmacokinetics of an Oral Contraceptive Pill When Coadministered to Healthy Female Volunteers
Brief Title: A Study of the Effects of GSK189075 on PK Profiles of an Oral Contraceptive Pill When Given to Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KG2107494
Record Dates: First submitted 2007-07-13; First posted 2007-07-20 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: healthy female,; pharmacokinetics,; pharmacodynamics; drug interaction,
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brevicon (Other): Oral contraceptive used to determine pharmacokinetics when given with GSK189075 to look for interaction.
  Interventions: Drug: GSK189075
- GSK189075 (Experimental): Given in conjunction with Brevicon to see if GSK189075 interfered with Brevicon drug levels.
  Interventions: Drug: Brevicon

INTERVENTIONS:
Drug: GSK189075 — Given with Brevicon to determine any effects of GSK189075 on Brevicon PK.
  Arms: Brevicon
Drug: Brevicon — Given with GSK189075 to determine if GSK189075 exerts an effect on GSK189075 PK.
  Other Names: GSK189075
  Arms: GSK189075

SUMMARY:
The purpose of this research study is to demonstrate a lack of effect of multiple doses of GSK189075 on the PK of an oral contraceptive pill in healthy female subjects. To estimate the effects of GSK189075 on hormonal levels and on birth control.

ELIGIBILITY:
Inclusion Criteria:

* healthy, non-smoking menstruating female age 18 to 45 years old, inclusive.
* able to take a specific oral contraceptive & KG2107494.
* female unable to have any more children, still has ovaries and uterus, and has a negative pregnancy test.
* female who can have children and who has regular periods and are willing to use an oral contraceptive pill and/or have a sterile partner.

Exclusion Criteria:

* pregnant or a nursing female.
* female subject able to have children of who is unwilling or unable to use an appropriate method of birth control at least 2 weeks prior to first dose of study drug until completion of the Follow-up visit.
* Have suffered with certain infection within 4 weeks prior to the first dose of study drug

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Oral contraceptive pill (OC) drug levels | over 24h starting on Day 14
blood hormone levels | on Days 1, 11-14, & 21 of Periods 1 (OC alone) & 3 (OC plus GSK study drug). Period 2 is GSK drug study alone.

SECONDARY OUTCOMES:
Adverse events | all visits after study drug
ECGs, Clinical laboratory tests | screening & follow-up
vital signs | screening;Day 13, Period 1 & 3; Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Miramar, Florida, United States